CLINICAL TRIAL: NCT07166094
Title: A Phase 3 Randomized, Open-label Study of Rinatabart Sesutecan (Rina-S) Versus Treatment of Investigator's Choice (IC) in Patients With Endometrial Cancer After Platinum-Based Chemotherapy and PD(L)-1 Therapy
Brief Title: Study to Assess the Efficacy and Safety of Rina-S Compared to Treatment of Investigator's Choice in Participants With Endometrial Cancer
Acronym: RAINFOL-03
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1184-03; jRCT2031250494 (Registry Identifier: Japan Registry for Clinical Trials (jRCT)); 2024-519818-31 (Other: EU CT Number); GOG-3128 (Other: Other Sponsor Identifier); ENGOT-en31 (Other: Other Sponsor Identifier); GEICO-158-E (Other: Other Sponsor Identifier)
Record Dates: First submitted 2025-09-09; First posted 2025-09-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer; Recurrent or Progressive Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rina-S (Experimental): Participants will receive Rina-S on Day 1 once every 3 weeks (Q3W).
  Interventions: Drug: Rina-S
- IC (Active Comparator): Participants will receive one of the following chemotherapies at the discretion of the investigator:
  * Paclitaxel on Days 1, 8, and 15 every 4 weeks (Q4W).
  * Doxorubicin on Day 1 Q3W.
  Interventions: Drug: IC

INTERVENTIONS:
Drug: Rina-S — Intravenous (IV) infusion.
  Other Names: Rinatabart Sesutecan; PRO1184; GEN1184
  Arms: Rina-S
Drug: IC — * Paclitaxel: IV infusion
  * Doxorubicin: IV bolus injection/infusion
  Arms: IC

SUMMARY:
The purpose of this study is to compare how well Rina-S (GEN1184) works compared to treatment of physician's choice (paclitaxel or doxorubicin) that are considered standard medical care for the treatment of recurrent or progressive endometrial cancer (EC) following prior therapy. There is an equal (50:50) chance of getting either Rina-S or a chemotherapy agent as treatment in this study.

The study duration will be approximately 3 years. The treatment duration will be different for every participant, but an average of 4 to 6 months is expected.

All participants will receive active drug; no one will be given placebo. Participation in the study will require visits to the study site(s).

DETAILED DESCRIPTION:
This is a global, open-label, randomized Phase 3 study in approximately 544 participants with recurrent or progressive EC following prior therapy.

Participants will be randomized in a 1:1 ratio to receive treatment with Rina-S vs investigator's choice (IC) (paclitaxel or doxorubicin). Investigators must select one of the IC treatment options for each participant prior to randomization so that this may be used for treatment assignment if the participant is randomized to the IC arm.

ELIGIBILITY:
Key Inclusion Criteria

* Participants must have histologically or cytologically confirmed recurrent or progressive endometrial cancer (EC; any subtype excluding neuroendocrine tumors, carcinosarcoma, or endometrial sarcoma) following prior therapy.
* Participants must have received at least 1, but not more than 3, prior lines of therapy:

  * Participants must have received prior platinum-based chemotherapy and a programmed death (ligand)-1 (PD(L)-1) inhibitor, either separately or in combination
  * If the tumor recurred more than 12 months after completion of platinum-based chemotherapy, additional platinum-based chemotherapy must be administered for recurrent disease unless the participant is ineligible for further platinum-based chemotherapy, in which case the reason for ineligibility must be documented.

    * Note: If Immunotherapy-based treatment is administered in the recurrent setting, then platinum rechallenge is not required, regardless of the duration of the platinum-free interval from prior platinum-based chemotherapy. In such cases, the reason for ineligibility for platinum-based chemotherapy must be documented.
  * Prior induction plus maintenance is considered 1 line of therapy
  * Hormonal therapy alone (ie, without chemotherapy) will not be counted as a separate line of therapy.
  * Therapy changed due to toxicity in the absence of progression will be considered part of the same line of therapy (i.e., will not be counted independently as a separate line of therapy)
* Participants must have progressed radiographically on or after their most recent line of therapy

Key Exclusion Criteria

* Prior therapy with an antibody-drug conjugate containing a topoisomerase 1 inhibitor.
* Has a past or current malignancy other than the inclusion diagnosis before the planned first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death (eg, 5-year OS ≥90%), including, but not limited to, adequately treated cervical carcinoma of Stage 1B or less, noninvasive basal cell or squamous cell skin carcinoma, noninvasive superficial bladder cancer, ductal carcinoma in situ, or any past malignancy considered cured for ≥3 years (ie, eligible participants must have complete response of ≥3 years duration).
* Known active central nervous system metastases or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry after completion of brain metastasis treatment, they have no new or enlarging brain metastases, and are off corticosteroids and anticonvulsants prescribed for symptoms associated with brain metastases for at least 7 days prior to the planned first dose of study drug. Participants with suspected brain metastases at screening should undergo a computed tomography (CT)/magnetic resonance imaging (MRI) of the brain prior to study entry.
* Hospitalization or clinical symptoms due to gastrointestinal obstruction within the past 91 days or radiographic evidence of gastrointestinal obstruction at the time of screening. Enrollment of participants who currently require parenteral nutrition must be discussed with the study medical monitor to determine eligibility.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per Response Criteria in Solid Tumors (RECIST) v1.1, as Determined by Investigator Assessment | Up to approximately 3 years
Overall Survival (OS) | Up to approximately 3 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR), per RECIST v1.1, as Determined by Investigator Assessment | Up to approximately 3 years
PFS, per RECIST v1.1, as Determined by Blinded Independent Central Review (BICR) | Up to approximately 3 years
ORR, per RECIST v1.1, as Determined by BICR | Up to approximately 3 years
Duration of Objective Response (DOR), per RECIST v1.1, as Determined by Investigator Assessment | Up to approximately 3 years
DOR, per RECIST v1.1, as Determined by BICR | Up to approximately 3 years
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 3 years
Change from Baseline in Global Health Status/Quality of Life (GHS/Qol) | Baseline up to approximately 3 years
Time to Deterioration (TTD) in GHS/Qol | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (15):
- United States (5):
  - Trials365, LLC, Shreveport, Louisiana
  - Sinai Hospital, Baltimore, Maryland
  - William Kahlert Reg. Can. Ctr, Westminster, Maryland
  - Willamette Valley Cancer Institute and Research Center - Eugene, Eugene, Oregon
  - USOR - Texas Oncology - Dallas Fort Worth (DFW), Fort Worth, Texas
- Japan (10):
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hyogo Cancer Center, Hyōgo
  - Niigata Cancer Center Hospital, Niigata
  - Saitama Medical University - International Medical Center, Saitama
  - Sapporo Medical University Hospital, Sapporo
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Cancer Institute Hospital of JFCR, Tokyo
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No